CLINICAL TRIAL: NCT06440694
Title: Colchicine to Quench the Inflammatory Response After Deep Vein Thrombosis: A Randomized Controlled Pilot Trial
Brief Title: Colchicine to Quench the Inflammatory Response After Deep Vein Thrombosis (The Conquer-DVT Pilot Trial)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONQUER-DVT Pilot
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism
Keywords: Proximal Lower Extremity Deep Vein Thrombosis; Randomized Trial; Colchicine; Post Thrombotic Syndrome; Inflammation
MeSH Terms: conditions — Venous Thromboembolism; Postthrombotic Syndrome; Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Pilot Trial comparing two groups - Colchicine 0.5 mg po once daily for 180 days vs Placebo 0.5 mg po once daily for 180 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Colchicine (Experimental): Colchicine 0.5 mg po once daily for 180 days. After the Day - 180 follow up, the study treatment will be discontinued and subsequent treatment will be at the discretion of the attending physician.
  Interventions: Drug: Colchicine 0.5 mg po
- Control Arm : Placebo (Placebo Comparator): Placebo 0.5 mg po once daily for 180 days. After the Day - 180 follow up, the study treatment will be discontinued and subsequent treatment will be at the discretion of the attending physician.
  Interventions: Drug: Placebo 0.5 mg po

INTERVENTIONS:
Drug: Colchicine 0.5 mg po — Colchicine 0.5 mg po once daily for 180 days.
  Other Names: Myinfla tablet 0.5 mg po daily
  Arms: Experimental Arm: Colchicine
Drug: Placebo 0.5 mg po — Placebo 0.5 mg po once daily for 180 days.
  Other Names: Placebo 0.5 mg po daily
  Arms: Control Arm : Placebo

SUMMARY:
This trial seeks to assess the feasibility of a full-scale, double-blind, placebo-controlled, randomized trial assessing whether low-dose colchicine (0.5 mg daily) reduces the risk of post-thrombotic syndrome (PTS) in patients with proximal lower extremity deep vein thrombosis (DVT).

DETAILED DESCRIPTION:
Eligible and consenting patients will be randomized via a central web-based randomization system (1:1 ratio) to receive one tablet of colchicine 0.5 mg or identical matching placebo daily starting within 7 days of initiation of anticoagulation for acute, symptomatic, proximal lower extremity Deep Vein Thrombosis (DVT) for a treatment course of 180 days (+/- 7 days). Study drug will start within 24 hours of randomization. The type, dose, and duration of anticoagulant therapy : unfractionated heparin, Low Molecular Weight Heparin (LMWH), fondaparinux, Direct Oral Anticoagulation (DOAC) or Vitamin K Agonist (VKA) will be left to the discretion of the treating physician or local investigator. The study drug will be continued until the end of the treatment period (180 days +/- 7 days). All patients will be observed until the end of study follow-up (365 days +/- 7 days).

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients 18 years of age or older with a first, acute, symptomatic proximal (popliteal vein or more proximal) objectively confirmed DVT of the lower extremity will be eligible to participate in the study.

Exclusion Criteria:

1. History of an allergic reaction or significant sensitivity to colchicine.
2. Requirement of colchicine for other indications.
3. Active or chronic diarrhea, or documented inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis), collagenous colitis or irritable bowel syndrome or existing blood dyscrasias.
4. Known or suspected, recent (<30 days) or active infections (acute or chronic).
5. History of cirrhosis, chronic active hepatitis, or severe liver disease.
6. Recent (<30 days) or chronic use of systemic (oral, intravenous) immunosuppressive drugs (including but not limited to steroids, tumor necrosis factor-alpha blockers, cyclosporine).
7. Known active cancer.
8. Any of the following as measured within the past 1-3 months or at screening: alanine, or aspartate aminotransferase >3 times the upper limit of normal, total bilirubin >2 times the upper limit of normal and a creatinine clearance by Cockcroft-Gault formula <30 mL/min.
9. Pregnancy, breast feeding or may be considering pregnancy during the study period or women of childbearing potential unwilling to use appropriate contraception during sex;
10. The use of medication with known drug-to-drug interactions (including but not limited to erythromycin or clarithromycin).
11. Unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pilot Trial Primary Outcome: Recruitment Rate | 12 months
  Mean number of participants recruited per site per month
Full-Scale Trial Primary Outcome: Post Thrombotic Syndrome | 180 days
  VILLALTA scale score ≥5 signifies clinically meaningful Post Thrombotic Syndrome

SECONDARY OUTCOMES:
Pilot Trial Secondary Outcome: Eligibility Rate | 12 months
  Proportion of screened patients who are eligible
Pilot Trial Secondary Outcome: Consent Rate | 12 months
  Proportion of eligible patients who provide consent
Pilot Trial Secondary Outcome: Retention Rate | 12 months
  Proportion of participants retained at follow-up
Pilot Trial Secondary Outcome: Study Completion Rate | 12 months
  Proportion of participants who completed all study procedures
Pilot Trial Secondary Outcome: Adherence Rate | 12 months
  Adherence to study drug measured by pill count at the end of follow-up
Pilot Trial Secondary Outcome: Reasons for declining participation | 12 months
  Pilot Trial Secondary Outcome: Reasons for declining participation
Full-Scale Trial Secondary Outcome: Post Thrombotic Syndrome | 365 days
  VILLALTA scale score ≥5 signifies clinically meaningful Post Thrombotic Syndrome
Full-Scale Trial Secondary Outcome: Severe Post Thrombotic Syndrome | 180 and 365 days
  VILLALTA scale score ≥ 15 signifies significant clinically meaningful Post Thrombotic Syndrome or presence of ulcer will be collected
Full-Scale Trial Secondary Outcome: Severity of Post Thrombotic Syndrome | 180 and 365 days
  Continuous VILLALTA score (VILLALTA scale score ≥5 signifies clinically meaningful Post Thrombotic Syndrome)
Full-Scale Trial Secondary Outcome: Patient Reported VILLALTA Scale | 180 and 365 days
  Full-Scale Trial Secondary Outcome: Patient Reported VILLALTA Scale (VILLALTA scale score ≥5 signifies clinically meaningful Post Thrombotic Syndrome)
Full-Scale Trial Secondary Outcome: Recurrent Venous Thromboembolism | 180 and 365 days
  Full-Scale Trial Secondary Outcome: Recurrent Venous Thromboembolism
Full-Scale Trial Secondary Outcome: Major Bleeding | 180 and 365 days
  As per International Society on Thrombosis and Haemostasis (ISTH) definition
Full-Scale Trial Secondary Outcome: Clinically Relevant Non-Major Bleeding | 180 and 365 days
  As per ISTH definition
Full-Scale Trial Secondary Outcome: Overall Mortality | 180 and 365 days
  Full-Scale Trial Secondary Outcome: Overall Mortality
Full-Scale Trial Secondary Outcome: Venous disease Specific Quality of Life | 180 and 365 days
  Scoring using VEINES-QOL/Sym (The VEINES-QOL summary score (based on 25 items) estimates the impact of chronic venous disease upon QOL)
Full-Scale Trial Secondary Outcome: Health-Related Quality of Life | 180 and 365 days
  Scoring using EuroQoL-EQ-5D-5L (EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state)
Full-Scale Trial Secondary Outcome: Incremental Cost-Effectiveness Ratio (ICER) | 180 and 365 days
  Full-Scale Trial Secondary Outcome: Incremental Cost-Effectiveness Ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Carrier, MD,MSc,FRCPC, Principal Investigator — Ottawa Hospital Research Institute / Division of Hematology- The Ottawa Hospital
Locations (3):
- Canada (3):
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Centre de recherche du Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - The Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
To be developed
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the full-scale trial
Access Criteria: Contact Principal Investigator